CLINICAL TRIAL: NCT06071780
Title: The Efficacy of Virgin Coconut Oil Contact Lens as Ocular Rewetting Agent on Dry Eyes
Brief Title: Virgin Coconut Oil Contact Lens as Ocular Rewetting Agent
Acronym: VCOCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Assoc Prof Dr Haliza Abdul Mutalib, Assoc Prof Dr, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: UKM1.21.3/244/NN-2019-042
Record Dates: First submitted 2023-09-16; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Dry Eyes
Keywords: Contact lens; VCO; TBUT; dry eyes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Both eyes of subjects will be instilled with either one of the study contact lens or the control lens at random.
Who Masked: Participant, Investigator
Masking Description: Only care provider was not masked as she had to insert the lens and to record the randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VCO contact lens (Active Comparator): contact lens soaked in VCO
  Interventions: Other: organic product - Virgin Coconut Oil
- control contact lens (Placebo Comparator): contact lens soaked in saline
  Interventions: Other: organic product - Virgin Coconut Oil

INTERVENTIONS:
Other: organic product - Virgin Coconut Oil — A commercially available sterilized contact lens was soaked in VCO for 4 hours in a sterile condition to allow absorption of VCO into the contact lens polymer. The contact lens here is a vehicle to transport the VCO into the eye.

SUMMARY:
This is a clinical trial where 44 subjects dry eyes were instilled with Virgin Coconut Oil (VCO CL) using contact lenses as its vehicle. All subjects are healthy subjects with no other ocular diseases except for having some dry eye symptoms (included with McMonnies questionnaires). Parameters measured at baseline and after 15 minutes of insertion and were compared. The control eyes were inserted with contact lenses soaked in saline (CCL). The eye that wears the VCO CL or the CCL were chosen randomly by masked operator. At the end of this study, the parameters measured will indicate if the VCO CL was able to retain tears in the eye and remove the dry eyes symptoms.

DETAILED DESCRIPTION:
A new study using contact lens pre-soaked in virgin coconut oil (VCO CL) was conducted to determine the safety of the agent on dry eye human. Efficacy of the VCO CL was assessed by measuring TBUT, anterior eye assessment, corneal staining, pH, and Schirmer value and the measurement of residual VCO volume in tears before instillation (0 minute) and at 15 minutes after insertion. Wilcoxon Signed Rank and Mann Whitney U Test were used to analyse any changes in all the measurable variables. The differences of the TBUT, corneal staining and residual VCO volume in tears value in both eyes were analyzed. These study data will suggest if the VCO CL is safe and effective and can be recommended to be used as an option for dry eyes in human

ELIGIBILITY:
Inclusion Criteria:

* Dry eye symptoms (according to McMonnies questionaires)
* Written consent

Exclusion Criteria:

* No ocular diseases
* No systemic diseases
* Not wearing contact lenses regularly for the past 6 months

Ages: 19 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
To compare the value of Tear Break-Up Time (TBUT) at baseline and 15 minutes after intervention | 15 minutes
  This is to evaluate the 'oil' component in the tearfilm
To compare the value of Schimer's Test at baseline and 15 minutes after intervention | 15 minutes
  This is to evaluate the aqueous component in the tear film
To compare the value of Corneal staining at baseline and 15 minutes after intervention | 15 minutes
  Fluorescein staining will indicate dry spots
To measure the oil stained area after intervention and to compare it with the control group | 15 minutes
  This oil stain will indicate the residual of VCO left in the eye after 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Haliza Abdul Mutalib, MOptom, Principal Investigator — National University of Malaysia
Locations (1):
- Optometry Clinic, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
when requested will be considered

REFERENCES:
- [Result] Mutalib HA, Kaur S, Ghazali AR, Chinn Hooi N, Safie NH. A pilot study: the efficacy of virgin coconut oil as ocular rewetting agent on rabbit eyes. Evid Based Complement Alternat Med. 2015;2015:135987. doi: 10.1155/2015/135987. Epub 2015 Feb 23. PMID 25802534

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT06071780/Prot_SAP_ICF_000.pdf